CLINICAL TRIAL: NCT02189408
Title: Effect of Platelet Rich Plasma ( PRP ) Applied During Knee Arthroscopy on Pain, Function and Quality of Life - A RCT With a Follow up of 12 Months
Brief Title: Clinical Study of Pain Reduction by Peri-arthroscopic PRP Application in Knee Degeneration
Acronym: PRP-Bochum
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Christian Duif MD, PostDoc Department of Orthopaedics, Ruhr University of Bochum
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRP-Bochum
Record Dates: First submitted 2014-06-11; First posted 2014-07-14 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2014-07

CONDITIONS: Knee Osteoarthritis; Cartilage Damage; Meniscal Tear
Keywords: Platelet rich plasma; Autologous conditioned plasma; Outerbridge
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PRP (Experimental): one intraoperative application of PRP in the interventional group
  Interventions: Biological: Platelet rich plasma
- Control (No Intervention): No application of any substance during knee arthroscopy

INTERVENTIONS:
Biological: Platelet rich plasma
  Other Names: ACP ( Arthrex )
  Arms: PRP

SUMMARY:
The purpose of this study is to investigate reduction of pain, gain of function and improvement of life quality by intraoperative applied platelet- rich- plasma ( PRP ) during knee arthroscopy for degeneration and osteoarthritis OA by conducting a randomized- controlled, double-blinded trial ( RCT ) including 58 patients with a follow up of 12 months and pain, assessed by Visual- Analogue Scale (VAS) after 6 months as primary endpoint.

ELIGIBILITY:
inclusion Criteria:

* degenerative knee pain
* age: > 18 years
* informed consent
* none to moderate comorbidity
* arthroscopy under general anaesthesia indicated

exclusion Criteria:

* trauma of the knee within the last 6 weeks before surgery
* circumscribed cartilage lesion with possibility of repair microfracture or autologous chondrocyte transplantation - procedures
* contraindications against PRP. application
* malignancies
* severe comorbidities
* age <18 years
* physically or mentally not able to provide informed consent
* severe knee instability
* corticosteroid injections within the last 6 weeks before surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2010-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
pain ( VAS ) | 6 months
  measurement of pain using a 100 mm VAS as platelet- rich-plasma demonstrated temporarily analgetic effects up to 6-9 months after application.

SECONDARY OUTCOMES:
pain ( VAS ) | 6 weeks, 12 months
  To investigate the pain development over the follow up period at the beginning and the end of our trial
knee function (Lysholm-score ) | 6 weeks, 6 months, 12 months
  to determine PRP-related gain of function according to time after application
quality of life ( physical und mental summaries of SF-36 German version ) | 6 weeks, 6 months and 12 months
  to identify a possible effect of PRP application on life quality ( physical and mental summaries )

CONTACTS AND LOCATIONS:
Overall Officials: Christoph von Schulze Pellengahr, MD, Study Director — Department of Orthopaedics, University Clinic of the Ruhr- University Bochum
Locations (1):
- Department of Orthopaedics at the St. Josef- Hospital, Bochum, Germany

REFERENCES:
- [Derived] Duif C, Vogel T, Topcuoglu F, Spyrou G, von Schulze Pellengahr C, Lahner M. Does intraoperative application of leukocyte-poor platelet-rich plasma during arthroscopy for knee degeneration affect postoperative pain, function and quality of life? A 12-month randomized controlled double-blind trial. Arch Orthop Trauma Surg. 2015 Jul;135(7):971-7. doi: 10.1007/s00402-015-2227-5. Epub 2015 May 10. PMID 25957981
- See also: Website of the Department of Orthopaedics — http://orthopaedie.klinikum-bochum.de/